CLINICAL TRIAL: NCT05999942
Title: A Gamma Scintigraphy Study to Investigate the Lung Deposition of Inhaled Amikacin-Loaded Liposomes in Healthy Male Volunteers
Brief Title: A Study to Investigate Lung Deposition of Inhaled Amikacin-loaded Liposomes in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD 201/23924
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Amikacin Liposome Inhalation (Experimental): Participants will receive a single dose of radiolabelled amikacin loaded liposomes by inhalation on Day 1.
  Interventions: Drug: Liposomal Amikacin for Inhalation

INTERVENTIONS:
Drug: Liposomal Amikacin for Inhalation — Administered via the Pari LC STAR™ nebulizer.
  Other Names: Amikacin Liposome Inhalation Suspension (ALIS),; Arikayce™

SUMMARY:
The primary purpose of this study is to determine the intra and extra pulmonary deposition and clearance of inhaled amikacin-loaded liposomes by gamma scintigraphy in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a body mass index (BMI) of 20-28.
* Participants with negative human immunodeficiency virus (HIV) and Hepatitis B and C results.
* Participants with no clinically significant findings in 12-lead electrocardiogram (ECG) determined within 14 days of the start of the study.

Exclusion Criteria:

* Participants who had clinically diagnosed asthma.
* Participants with a known allergic reaction to amikacin, liposomes or any of the radiolabelling products (i.e. [^99m]Tc, or [^111]In, and [^81m]Kr).
* Evidence of clinically significant pulmonary, renal, hepatic, cardiovascular or metabolic dysfunction.
* History of smoking within the past 12 months.
* History of chronic cough or wheezing within the previous 21 days.
* Participants who had an upper respiratory illness or infection within the previous 21 days.
* A history of drug or alcohol abuse.
* Donation of 450 milliliters (mL) or more blood within the previous 12 weeks.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2004-06-02 (Actual); Primary Completion 2004-06-29 (Actual); Study Completion 2004-06-29 (Actual)

PRIMARY OUTCOMES:
Pulmonary Deposition of Radiolabelled Amikacin-loaded Liposomes Measured as Percentage Retention of Emitted Dose Deposited in the Lungs | Pre-administration and 2 hours post-administration on Day 1

SECONDARY OUTCOMES:
Percent Dose Deposited in Oropharyngeal and Stomach Region | At multiple timepoints post-administration up to Day 2
Percent Dose Remaining in the Device Including the Mouthpiece | At multiple timepoints post-administration up to Day 2
Percent Dose Remaining in the Low Resistance Exhalation Filter | At multiple timepoints post-administration up to Day 2
Penetration Index Based on the Ratio of Counts in the Central:Peripheral Lung Regions, Corrected for Regional Lung Volume (sC/P) | Pre-administration and 2 hours post- administration on Day 1

IPD SHARING:
Plan to Share IPD: No